CLINICAL TRIAL: NCT03501472
Title: Pictorial Warning Labels, Numeracy, and Memory for Numeric Cigarette Health-risk Information Over Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ellen Peters, Professor, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: P50CA180908A2b; P50CA180908 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Smoking, Cigarette; Smoking Cessation
Keywords: pictorial warning labels; risk knowledge; emotion; memory; risk perceptions; quit intentions; numeracy
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Text-only PWL, immediate post (Experimental): Exposure to 4 FDA-mandated warning labels and numeric risk information for 8 outcomes related to those warnings (2 outcomes for each PWL; half as percentage, half as frequency)
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered immediately following last exposure to warning labels
  Interventions: Behavioral: text-only PWL; Behavioral: immed posttest
- Text-only PWL, delay posttest (Experimental): Exposure to 4 FDA-mandated warning labels and numeric risk information for 8 outcomes related to those warnings (2 outcomes for each PWL; half as percentage, half as frequency)
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered 6 weeks following last exposure to warning labels
  Interventions: Behavioral: text-only PWL; Behavioral: delay posttest
- Low-emot PWL, immed post (Experimental): Exposure to 4 FDA-mandated warning labels paired with images that elicit little emotion and numeric risk information for 8 outcomes related to those warnings (2 outcomes for each PWL; half as percentage, half as frequency)
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered immediately following last exposure to warning labels
  Interventions: Behavioral: low-emot PWL; Behavioral: immed posttest
- Low-emot PWL, delay posttest (Experimental): Exposure to 4 FDA-mandated warning labels paired with images that elicit little emotion and numeric risk information for 8 outcomes related to those warnings (2 outcomes for each PWL; half as percentage, half as frequency)
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered 6 weeks following last exposure to warning labels
  Interventions: Behavioral: low-emot PWL; Behavioral: delay posttest
- High-emot PWL, immed posttest (Experimental): Exposure to 4 FDA-mandated warning labels paired with images that elicit high emotion and numeric risk information for 8 outcomes related to those warnings (2 outcomes for each PWL; half as percentage, half as frequency)
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered immediately following last exposure to warning labels
  Interventions: Behavioral: high-emot PWL; Behavioral: immed posttest
- High-emot PWL, delay posttest (Experimental): Exposure to 4 FDA-mandated warning labels paired with images that elicit high emotion and numeric risk information for 8 outcomes related to those warnings (2 outcomes for each PWL; half as percentage, half as frequency)
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered 6 weeks following last exposure to warning labels
  Interventions: Behavioral: high-emot PWL; Behavioral: delay posttest

INTERVENTIONS:
Behavioral: text-only PWL
  Arms: Text-only PWL, delay posttest; Text-only PWL, immediate post
Behavioral: low-emot PWL
  Arms: Low-emot PWL, delay posttest; Low-emot PWL, immed post
Behavioral: high-emot PWL
  Arms: High-emot PWL, delay posttest; High-emot PWL, immed posttest
Behavioral: immed posttest
  Arms: High-emot PWL, immed posttest; Low-emot PWL, immed post; Text-only PWL, immediate post
Behavioral: delay posttest
  Arms: High-emot PWL, delay posttest; Low-emot PWL, delay posttest; Text-only PWL, delay posttest

SUMMARY:
Pictorial cigarette warning labels (PWLs) are thought to increase risk knowledge, but experimental research has not examined PWLs' longer term effects on memory for health risks, or for numeric risks (e.g., percentage risk for developing lung cancer). This trial tests memory for numeric health risks immediately or after a six-week delay for US adult smokers. In addition, the trial tests the effects of different warning label components (e.g., whether the numeric risks are percentage or frequency), participants' level of numeric ability, and the consequences of memory for numeric risks on participant risk perceptions and quit intentions.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* have smoked 100+ lifetime cigarettes
* currently smoke "every day" or "some days."
* US resident

Exclusion Criteria:

* have not ever smoked a cigarette

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2016-04-16 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
numeric risk recall | immediately following last exposure or after 6-week delay
  free recall for numeric risks presented in labels (e.g., ____% of smokers die before age 85), both for smokers and nonsmokers
numeric risk recognition | immediately following last exposure or after 6-week delay
  Participants answered one multiple choice question about the numeric risk for smokers and nonsmokers (combined in one question) for each of the 8 outcomes that had been paired with the PWLs. For each question, there were four decoy responses.

SECONDARY OUTCOMES:
smoking risk perceptions | immediately following last exposure or after 6-week delay
  Participants completed several scale items about how much risk they perceived smoking posed to them (e.g., "Compared to the average nonsmoker your age, gender, and race, how would you rate your chances of": 1) "getting a life threatening illness because of smoking," 2) "getting lung cancer," and 3) "dying at a younger age than average" (-3 = Much lower, +3 = Much higher))
  They also gave verbal likelihood ratings for each of the 8 outcomes of smoking that had been paired with the labels (e.g., "Thinking of risks that you were shown in the warnings, what is the likelihood of a smoker [non-smoker] dying from heart disease?," 0=impossible, 11=certain)
smoking risk knowledge | immediately following last exposure or after 6-week delay
  Participants listed as many risks of smoking as they could think of.
quit intentions | immediately following last exposure or after 6-week delay
  Participants intentions to quit smoking, Likelihood of smoking within next 30 days, next year (-3 = very unlikely, 3 = very likely)